CLINICAL TRIAL: NCT01402882
Title: Tranexamic Acid for the Treatment of Significant Traumatic Brain Injury: an International Randomised, Double Blind Placebo Controlled Trial
Brief Title: Clinical Randomisation of an Antifibrinolytic in Significant Head Injury
Acronym: CRASH-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISRCTN15088122
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2018-03

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; tranexamic acid; antifibrinolytic; randomised; clinical trial
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Experimental)
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): (Sodium Chloride 0.9%)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 2 grams (1 gram over 10 minutes and 1 gram over 8 hours)

SUMMARY:
The CRASH-3 trial will provide reliable evidence about the effect of tranexamic acid on mortality and disability in patients with traumatic brain injury. The effect of tranexamic acid on the risk of vascular occlusive events and seizures will also be assessed. Additionally, a nested study will be conducted in a subset of CRASH-3 trial participants. This nested study (CRASH-3 Intracranial Bleeding Sub-Study [CRASH-3 IBS]) will examine the effect of tranexamic acid on intracranial haemorrhage and cerebral ischaemia using CT Scans in approximately 1,000 patients randomised into the CRASH-3 trial.

DETAILED DESCRIPTION:
BACKGROUND: Worldwide, over 10 million people are killed or hospitalised because of traumatic brain injury (TBI) each year. About 90% of deaths from TBI occur in low and middle income countries. TBI mostly affects young adults and many experiencing long lasting or permanent disability. The social and economic burden of TBI is considerable. Tranexamic acid (TXA) is commonly given to surgical patients to reduce bleeding and the need for blood transfusion. TXA has been shown to reduce the number of patients receiving a blood transfusion by about a third, reduces the volume of blood transfused by about one unit, and halves the need for further surgery to control bleeding in elective surgical patients. More recently, the CRASH-2 trial showed that the administration of TXA within 8 hours of injury significantly reduces deaths due to bleeding (RR=0.85, 95% CI 0.76-0.96; p=0.008), and all-cause mortality (RR=0.91, 95% CI 0.85-0.97; p=0.0035), with no apparent increase in vascular occlusive events. A meta-analysis of randomised controlled trials of TXA in TBI showed a significant reduction in haemorrhage growth (OR=0.61, 95%CI 0.41 to 0.91) and mortality (OR=0.59, 95%CI 0.35 to 0.99) with TXA. Although the results from these trials are promising, the estimates are imprecise and there are no data on the effect of TXA on disability. Additionally, a nested study will be conducted in a subset of CRASH-3 trial participants. This nested study (CRASH-3 Intracranial Bleeding Sub-Study [CRASH-3 IBS]) will examine the effect of tranexamic acid on intracranial haemorrhage and cerebral ischaemia using CT Scans in approximately 1,000 patients randomised into the CRASH-3 trial.

AIM: The CRASH-3 trial will provide reliable evidence about the effect of tranexamic acid on mortality and disability in patients with TBI. The effect of TXA on the risk of vascular occlusive events and seizures will also be assessed.

PRIMARY OUTCOME: The primary outcome is death in hospital (within 28 days of injury) of patients randomised within 3 hours of injury (cause of death will be described).

SECONDARY OUTCOMES:

1. Vascular occlusive events (myocardial infarction, stroke, pulmonary embolism, clinical evidence of deep vein thrombosis)
2. In hospital disability assessed using the Disability Rating Scale and Patient Orientated Outcome
3. Seizures
4. Neurosurgical intervention
5. Days in intensive care Other adverse events will be described

Other Outcome Measures: CRASH-3 IBS Primary outcome - the total volume of intracranial haemorrhage after randomisation, adjusting for baseline haemorrhage volume.

Secondary outcome -

* Frequency of progressive haemorrhage: number of patients with a post-randomisation CT scan with total haemorrhage volume of more than 25% of the volume on the pre-randomisation scan;
* Frequency of delayed haemorrhage: number of patients with haemorrhage on the post-randomisation CT scan when there was not one on the pre-randomisation scan;
* New focal ischaemic lesions: ischaemic lesions which appear on the post-randomisation CT scan but not on the pre-randomisation scan;
* Total volume of intracranial bleeding in patients who undergo surgical evacuation of haemorrhage after randomisation, adjusting for volume of baseline bleeding.

TRIAL DESIGN: A large, pragmatic, randomised, double blind, placebo controlled trial among 13,000 traumatic brain injury patients

DIAGNOSIS AND INCLUSION/EXCLUSION CRITERIA:

Adults with traumatic brain injury who

* are within eight hours of injury
* with any intracranial bleeding on CT scan or who have a GCS of 12 or less, and
* have no significant extra-cranial haemorrhage The fundamental eligibility criterion is the responsible clinician's 'uncertainty' as to whether or not to use tranexamic acid in a particular patient with traumatic brain injury.

TEST PRODUCT, REFERENCE THERAPY, DOSE AND MODE OF ADMINISTRATION: A loading dose of tranexamic acid

(1 gram by intravenous injection) or placebo (sodium chloride 0.9%) will be given as soon as possible after randomisation. A maintenance dose of tranexamic acid (1 gram by intravenous injection) or placebo (sodium chloride 0.9%) will be given after the loading dose is finished.

SETTING: This trial will be coordinated from the London School of Hygiene & Tropical Medicine (University of London) and conducted worldwide in hospitals in low, middle and high income countries.

ELIGIBILITY:
Inclusion Criteria:

Adults with traumatic brain injury who

* are within eight hours of injury (limited to within 3 hours from September, 2016)
* with any intracranial bleeding on CT scan or who have a GCS of 12 or less, and
* have no significant extra-cranial haemorrhage The fundamental eligibility criterion is the responsible clinician's 'uncertainty' as to whether or not to use tranexamic acid in a particular patient with traumatic brain injury

Exclusion Criteria:

The fundamental eligibility criterion is the responsible clinician's 'uncertainty' as to whether or not to use tranexamic acid in a particular patient with traumatic brain injury

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12737 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is death in hospital in patients recruited within 3 hours and cause of death will be described. | within 28 days of injury

SECONDARY OUTCOMES:
(a) Vascular occlusive events (myocardial infarction, stroke, pulmonary embolism, clinical evidence of deep vein thrombosis) | Prior death, discharge or 28 days
(b) In hospital disability assessed using the Disability Rating Scale and Patient Orientated Outcome | Prior death, discharge or 28 days
(c) Seizures | Prior death, discharge or day 28
(d) Neurosurgical intervention | prior death, discharge or day 28
(e) Days in intensive care | prior death, discharge or day 28
(f) Other adverse events | prior death, discharge or day 28

OTHER OUTCOMES:
CRASH-3 IBS: Primary outcome - the total volume of intracranial haemorrhage | 1) CT scan done before receipt of trial treatment; (2) CT scan done after receipt of trial treatment (up to 28 days after randomisation)
Frequency of progressive haemorrhage: number of patients with a post-randomisation CT scan with total haemorrhage volume of more than 25% of the volume on the pre-randomisation scan | 1) CT scan done before receipt of trial treatment; (2) CT scan done after receipt of trial treatment (up to 28 days after randomisation)
Frequency of delayed haemorrhage: | 1) CT scan done before receipt of trial treatment; (2) CT scan done after receipt of trial treatment (up to 28 days after randomisation)
New focal ischaemic lesions: | 1) CT scan done before receipt of trial treatment; (2) CT scan done after receipt of trial treatment (up to 28 days after randomisation)
• Total volume of intracranial bleeding in patients who undergo surgical evacuation of haemorrhage after randomisation | 1) CT scan done before receipt of trial treatment; (2) CT scan done after receipt of trial treatment (up to 28 days after randomisation)

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Shakur, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- High Technology Medical Center, University Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Yes
After all relevant publications are completed, totally anonymised data will be available at https://ctu-app.lshtm.ac.uk/freebird/

REFERENCES:
- [Derived] Mansukhani R, Belli A, Brenner A, Chaudhri R, Frimley L, Faizah Jamaluddin S, Jooma R, Shakur-Still H, Shokunbi T, Roberts I. Effect of early tranexamic acid treatment on fatigue in patients with mild traumatic brain injury: data from the CRASH-3 clinical trial. Wellcome Open Res. 2024 Oct 28;6:346. doi: 10.12688/wellcomeopenres.17421.3. eCollection 2021. PMID 39502454
- [Derived] Roberts I, Shakur-Still H, Aeron-Thomas A, Beaumont D, Belli A, Brenner A, Cargill M, Chaudhri R, Douglas N, Frimley L, Gilliam C, Geer A, Jamal Z, Jooma R, Mansukhani R, Miners A, Pott J, Prowse D, Shokunbi T, Williams J. Tranexamic acid to reduce head injury death in people with traumatic brain injury: the CRASH-3 international RCT. Health Technol Assess. 2021 Apr;25(26):1-76. doi: 10.3310/hta25260. PMID 33928903
- [Derived] Brenner A, Belli A, Chaudhri R, Coats T, Frimley L, Jamaluddin SF, Jooma R, Mansukhani R, Sandercock P, Shakur-Still H, Shokunbi T, Roberts I; CRASH-3 trial collaborators. Understanding the neuroprotective effect of tranexamic acid: an exploratory analysis of the CRASH-3 randomised trial. Crit Care. 2020 Nov 11;24(1):560. doi: 10.1186/s13054-020-03243-4. PMID 33172504
- [Derived] Mansukhani R, Frimley L, Shakur-Still H, Sharples L, Roberts I. Accuracy of time to treatment estimates in the CRASH-3 clinical trial: impact on the trial results. Trials. 2020 Jul 25;21(1):681. doi: 10.1186/s13063-020-04623-5. PMID 32711551
- [Derived] CRASH-3 trial collaborators. Effects of tranexamic acid on death, disability, vascular occlusive events and other morbidities in patients with acute traumatic brain injury (CRASH-3): a randomised, placebo-controlled trial. Lancet. 2019 Nov 9;394(10210):1713-1723. doi: 10.1016/S0140-6736(19)32233-0. Epub 2019 Oct 14. PMID 31623894
- [Derived] Roberts I, Belli A, Brenner A, Chaudhri R, Fawole B, Harris T, Jooma R, Mahmood A, Shokunbi T, Shakur H; CRASH-3 trial collaborators. Tranexamic acid for significant traumatic brain injury (The CRASH-3 trial): Statistical analysis plan for an international, randomised, double-blind, placebo-controlled trial. Wellcome Open Res. 2018 Sep 26;3:86. doi: 10.12688/wellcomeopenres.14700.2. eCollection 2018. PMID 30175246
- [Derived] Mahmood A, Roberts I, Shakur H. A nested mechanistic sub-study into the effect of tranexamic acid versus placebo on intracranial haemorrhage and cerebral ischaemia in isolated traumatic brain injury: study protocol for a randomised controlled trial (CRASH-3 Trial Intracranial Bleeding Mechanistic Sub-Study [CRASH-3 IBMS]). Trials. 2017 Jul 17;18(1):330. doi: 10.1186/s13063-017-2073-6. PMID 28716153
- [Derived] Dewan Y, Komolafe EO, Mejia-Mantilla JH, Perel P, Roberts I, Shakur H; CRASH-3 Collaborators. CRASH-3 - tranexamic acid for the treatment of significant traumatic brain injury: study protocol for an international randomized, double-blind, placebo-controlled trial. Trials. 2012 Jun 21;13:87. doi: 10.1186/1745-6215-13-87. PMID 22721545
- See also: Trial website — http://crash3.lshtm.ac.uk/